CLINICAL TRIAL: NCT02832973
Title: Resistant Hypertension On Treatment - Sequential Nephron Blockade Compared to Dual Blockade of the Renin-angiotensin-aldosterone System Plus Bisoprolol in the Treatment of Resistant Arterial Hypertension: A Randomized Trial (ResHypOT)
Brief Title: Sequential Nephron Blockade vs. Dual Blockade Renin-angiotensin System + Bisoprolol in Resistant Arterial Hypertension
Acronym: ResHypOT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sao Jose do Rio Preto Medical School (Other)
Responsible Party: Principal Investigator, Juan Carlos Yugar Toledo, MD, PhD, Sao Jose do Rio Preto Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SaoJoseRPU
Record Dates: First submitted 2016-06-12; First posted 2016-07-14 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Hypertension Resistant to Conventional Therapy
Keywords: Hypertension Resistant to Conventional Therapy; Natriuretic Agents; Renin-Angiotensin System; Bisoprolol
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy | interventions — Spironolactone; Furosemide; Amiloride; Ramipril; Angiotensin-Converting Enzyme Inhibitors; Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spironolactone, Furosemide Amiloride (Experimental): Spironolactone 25 mg qd, Furosemide 20 mg qd, Furosemide 40 mg qd, Amiloride 5 mg qd
  Interventions: Drug: Spironolactone; Drug: Furosemide,; Drug: Amiloride
- Ramipril, Bisoprolol (Active Comparator): Ramipril 5 mg qd, Ramipril 10 mg qd, Bisoprolol 5 mg qd, Bisoprolol 10 mg qd
  Interventions: Drug: Ramipril; Drug: Bisoprolol

INTERVENTIONS:
Drug: Spironolactone — Spironolactone 25 mg
  Other Names: Natriuretic diuretics
  Arms: Spironolactone, Furosemide Amiloride
Drug: Furosemide, — Furosemide 20-40 mg
  Other Names: Furosemide 20-40 mg
  Arms: Spironolactone, Furosemide Amiloride
Drug: Amiloride — Amiloride 5 mg
  Other Names: Amiloride 5 mg
  Arms: Spironolactone, Furosemide Amiloride
Drug: Ramipril — Ramipril 5-10 mg
  Other Names: ACE inhibitor
  Arms: Ramipril, Bisoprolol
Drug: Bisoprolol — Bisoprolol 5-10 mg
  Other Names: Betablocker
  Arms: Ramipril, Bisoprolol

SUMMARY:
A randomized clinical trial comparing sequential nephron blockage (SNB) with dual blockade of the renin-angiotensin system (RAAS) plus bisoprolol (DBB) in the treatment of resistant arterial hypertension (RH) was designed to investigate the importance of the SNB and the contribution of its volume component versus DBB and the importance of the serum renin in maintaining BP levels. This randomized trial with two treatment arms could help tailor therapy by identifying a more effective choice to control hypertension whether by acting on the control of volume or sodium balance, or by acting on the effects of the RAAS on the kidney.

Methods - Participants: 80 patients undergoing treatment for RH with losartan (100-200 mg), chlorthalidone (25 mg), and amlodipine (5 mg) will be randomly divided into two groups after applying inclusion and exclusion criteria.

Group 1: Sequential nephron blockade (SNB Group) n = 40 Group 2: Dual blockade of the RAAS plus bisoprolol (DBB Group) n = 40 Intervention: SNB consists in a progressive increase in sodium depletion. After the administration of a thiazide diuretic (chlorthalidone) and aldosterone receptor blocker, low doses of furosemide are administered and subsequently amiloride is prescribed to enhance the natriuretic effect.

The dual blockade of the RAAS plus bisoprolol is used to increase the effect of angiotensin receptor 1 blockers (ARBs). Therapy then requires sequentially adding an angiotensin converting enzyme (ACE) inhibitor to reduce the levels of angiotensin (Ang) II resulting from blockage of the Ang II receptor and then to administer a beta-blocker to decrease the elevated renin secretion due to both the ACE inhibitors and ARBs Objective: This study, which compares two antihypertensive treatment regimens in patients with RH, has the following objectives: to demonstrate the therapeutic efficacy of SNB against DBB in RH patients, and to assess the side effects and adherence to treatment over 20 weeks of treatment.

Enrollment: The eligibility criteria will follow those shown in the flowchart for the diagnosis of RH of the First Brazilian Position on RH.

Patients will be excluded if they have: chronic renal failure, atrial fibrillation/atrioventricular block, contraindication to the drugs that will be used, refusal or failure to follow the regimen and secondary hypertension.

Follow-up: Patients will be analyzed in five visits at intervals of 28 days for 20 weeks

DETAILED DESCRIPTION:
Introduction

Resistant hypertension (RH) is characterized when the blood pressure (BP) remains above the recommended goal after taking three antihypertensive drugs with synergistic actions, at their maximum recommended tolerated doses for at least six months; one preferably should be a diuretic. True RH should be differentiated from pseudo resistance, which occurs due to non-adherence to treatment, inadequate BP measurements, inadequate doses of medications, inappropriate therapeutic regimens, or the presence of the so-called white-coat effect.

The exact prevalence of RH is unknown. In controlled randomized studies with thousands of hypertensive patients, approximately 25% to 30% of participants did not achieve the BP goal recommended by guidelines despite receiving three or more antihypertensive drugs; these studies included careful assessments of adherence to therapy and even ambulatory BP monitoring (ABPM), which excludes patients with pseudo resistance.

Observational data from the North American National Health and Nutrition Examination Survey (NHANES) collected in 2003-2008 showed that the prevalence of RH among adults diagnosed with hypertension (HTN) in this period was 8.9% and among adults on antihypertensive treatment, it was 12.8%. Similarly, a large population study in Spain (68,000 patients) found that the prevalence of RH was 14.8% among those treated for HTN. Based on these recent studies, it is justifiable to say that the prevalence of RH is about 14%. RH is a difficult-to-manage clinical condition due to failure of patients to adhere to treatment, the physician's difficulty to adjust the medication because of genetic factors that hinder the effectiveness of treatment and medical inertia.

Pathophysiology of resistant hypertension: The mechanisms involved in the pathophysiology of RH are the vascular smooth muscle tone and increased blood volume, intensification of the activity of the sympathetic system and hyperactivity of the renin-angiotensin-aldosterone system (RAAS). Increased sensitivity to sodium appears to be the main factor in understanding the pathophysiology of this syndrome, not only as it incorporates the above mechanisms, but also as it explains, in part, the variability of therapeutic response of patients with RH. The RAAS is vital to the regulatory system that controls total body sodium as are atrial natriuretic peptide factors and pressure receptors in the atria and kidney. Sodium and water retention can lead to resistance against antihypertensive drugs. Under the physiological point of view, BP is maintained by continuous regulation of cardiac output and peripheral vascular resistance exerted at three anatomic sites: arterioles, postcapillary venules (capacitance vessels) and the heart. A fourth anatomical site of control, the kidney, contributes to the maintenance of BP by regulating intravascular volume.

Rational:

Thus, identifying the contribution of volume and serum renin in maintaining BP levels could help tailor treatment with a more effective choice for hypertension control, whether by acting on the control of volume or sodium balance, or by acting on the effects of the RAAS on the kidney.

Sequential nephron blockade consists in a progressive increase in sodium depletion. After the administration of a thiazide diuretic (chlorthalidone) and aldosterone receptor blocker, low doses of furosemide are administered and subsequently amiloride is prescribed to enhance the natriuretic effect.

The blockade of the RAAS is to increase the effect of the angiotensin receptor 1 blockers (ARBs). Therapy then requires sequentially adding an angiotensin converting enzyme (ACE) inhibitor to reduce the levels of angiotensin (Ang) II resulting from the blockage of the Ang II receptor and then to administer a beta-blocker to decrease the elevated renin secretion due to both the ACE inhibitors and ARBs.

Research question:

The following research questions will be explored: Do sequential nephron blockade (SNB) and dual blockade of the renin-angiotensin-aldosterone system plus bisoprolol (DBB) constitute good therapeutic options in the reduction of peripheral blood pressure of patients with RH? Which therapeutic option is able to reduce the central BP of resistant hypertensive patients? Is the strategy of SNB as good as DBB? Objectives: This study will compare two antihypertensive treatment regimens in RH patients of the Medical School in Sao Jose do Rio Preto. It aims to demonstrate the therapeutic efficacy of SNB against DBB in RH patients, and to assess the side effects, and adherence to therapy over 20 weeks of treatment.

Methods:

A randomized clinical trial with two therapeutic regimens for RH, SNB and DBB, will be compared in an open-label prospective study at the Medical School in Sao Jose do Rio Preto.

Eighty patients undergoing treatment for RH with losartan (100-200 mg), chlorthalidone (25 mg), and amlodipine (5 mg) will be randomly divided into two groups after applying inclusion and exclusion criteria.

Group 1: Sequential nephron blockade (SNB Group) - 40 patients will receive in addition to the basal therapy, spironolactone (25 mg), spironolactone 25 mg plus furosemide (20 mg), spironolactone (25 mg) plus furosemide (40 mg) and spironolactone (25 mg) plus furosemide (40 mg) plus amiloride (5 mg), sequentially.

Group 2: Dual blockade of the renin-angiotensin-aldosterone system plus bisoprolol (DBB Group) - 40 patients will receive, in addition to the basal therapy, ramipril (5 mg), ramipril (10 mg), ramipril (10 mg) plus bisoprolol (5 mg) and ramipril (10 mg) plus bisoprolol (10 mg), sequentially.

Forty patients fulfilling the following criteria will be enrolled in each group:

The project was approved by the Research Ethics Committee of Hospital de Base of the Medical School in São José do Rio Preto (FAMERP) and Brazilian Research Ethics Committee (# 33943014.6.0000.5415).

The nature of the study was carefully explained to patients and all individuals, after agreeing to participate in the study, signed informed consent forms and filled out a standard questionnaire.

Measurement of BP including 24-h ambulatory BP monitoring (ABPM): The BP will be measured by the indirect method, following the VI Brazilian Guidelines for the Treatment of Hypertension.

ABPM and home BP measurement will be carried out as additional tools to investigate hypertension according to the technical norms of the 5th Brazilian Guidelines on Ambulatory Blood Pressure Monitoring.

ABPM will be performed using the Mobil-O-Graph (Netherlands). Anthropometric measurements (Weight and height), measured by anthropometric scales, will be used to calculate the body mass index (BMI) utilizing the formula BMI = weight (kg)/height squared (m²). The abdominal circumference will be measured at the midpoint between the iliac crest and the lower costal margin. Values equal to or below 80 cm and 94 cm are considered appropriate for women and for men, respectively.

Biochemical tests and imaging: Blood samples will be drawn from all patients at the first and last visits after fasting for 12 hours to measure total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, very low-density lipoprotein cholesterol, triglycerides, glucose, insulin, creatinine, sodium and potassium.

All patients will be submitted to electrocardiography, echocardiography, carotid Doppler, ultrasound with Doppler of the renal arteries, stress testing and radial artery applanation tonometry (AT).

Study design:

Patients will be analyzed in five visits at 28-day intervals. V zero: Week -4 to Week 0. All patients will remain under treatment with losartan (100 - 200 mg), chlorthalidone (25 mg), and amlodipine (5 mg). Individuals with BP > 135/85 mmHg by ABPM will be randomized to one of the study groups.

V1: Week 0 to Week 4. Individuals receive 25 mg of spironolactone (SNB Group) or 5 mg of ramipril (DBB Group).

V2: Week 4 to Week 8. Individuals with BP <135/85 mmHg by ABPM will continue using the same regimen. Subjects with BP >135/85 mmHg by ABPM will receive in addition to their existing regimen, furosemide (20 mg) for the SNB Group and ramipril (10 mg) for the DBB Group.

V3: Week 8 to Week 12. Subjects with BP <135/85 mmHg by ABPM will continue on the same regimen. Individuals with BP >135/85 mmHg by ABPM will receive an extra 40 mg of furosemide for patients in the SNB Group and 5 mg of bisoprolol for patients in the DBB Group.

V4: Week 12 to Week 16. Subjects with BP <135/85 mmHg by ABPM will continue using the same regimen. Individuals with BP >135/85 mmHg by ABPM will receive an extra 5 mg of amiloride for patients in the SNB Group and 10 mg of bisoprolol for patients in the DBB Group.

V5: Week 16 to Week 20. Subjects will continue using the same regimen. Blood samples will be drawn from all patients. Radial artery applanation tonometry and ABPM will be performed.

Statistical analysis The t-test or Wilcoxon test for quantitative variables and chi-square and Fisher test for qualitative variables were used in the comparative analysis of the clinical characteristics of RHTN patients. Data were expressed as means ± 1 standard deviation.

The sample size was estimated at 72 individuals for an expected zero difference with a SD of 12 mmHg to demonstrate the non-inferiority of the strategy of SNB compared to RASDB plus bisoprolol assuming an absolute difference of ≤ 5 mmHg for systolic BP.

Non-inferiority was evaluated for a one-sided 95% confidence interval (CI) estimated by a linear mixed model for repeated measures. P-values <0.05 will be considered statistically significant.

Primary outcomes:

Reduction of systolic BP, diastolic BP, mean BP and pulse pressure after 20 weeks of treatment with sequential nephron blockade compared to dual blockade of the renin-angiotensin-aldosterone system plus bisoprolol.

Secondary outcomes:

Safety and tolerability, biochemical changes, evaluation of the renal function and recognition of hypotension (ABPM). Assessment of BP outcomes (mean of three measurements by an automatic electronic device - Omron 711) and hemodynamic parameters (Omron 9000 device) will be measured in the office at all follow-up visits.

Missing or dropout Participants: Patients will be registered with a phone number and address for further contact in case of missing visits.

Sample size:

The calculation of the sample size with an alpha error of 5%, statistical power of 80%, standard deviation of 8 mmHg, and maximum acceptable absolute difference of 6 mmHg (diastolic BP), indicated the necessity to study 36 patients per group (SNB versus DBB). However, considering a potential rate of 10-15% dropout or loss to follow-up, 40 will be considered for each group. The difference of 5 mmHg (diastolic BP) has been achieved, on average, in clinical trials that have demonstrated the advantage of one drug over placebo or other non-pharmacological treatments in the prevention of major cardiovascular outcomes.

No washout period will be used. Results Baseline clinical characteristics and laboratory parameters of the 72 patients with primary resistant hypertension randomized to SNB (n=35) or RASDB (n=37) were similar across both study groups. At the end of the study, a significant reduction of the office pressure was observed (SBP and DBP) in both after intervention groups SNB group: initial SBP: 174.5 ± 21.08; final SBP: 127.0 ± 14.74; Initial DBP: 105.3 ± 15.5, final DBP: 78.11 ± 9.28 (p <0.0001), RASDB group: initial SBP: 178.4 ± 21.08, final SBP: 134.4 ± 23.25, initial DBP: 102.7 ± 11.07, final DBP: 77.33 ± 13.75 (p <0.0001).

Central systolic pressure had a greater reduction in the SNB group (p <0.005). ABPM had a significant reduction of SBP and DBP in both groups (SNB group p <0.0001 for SBP and DBP before x after intervention, RASDB group p <0.0001 for SBP and DBP before x after intervention). No discontinuation due to drug-related adverse events in both study groups.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Resistant Hypertension Must to able swallow antihypertensive drug classes at maximum tolerated doses.

.

Exclusion Criteria:

Secondary Hypertension Chronic renal failure Coronary artery disease Atrial fibrillation Atrioventricular block Refuse or fail to follow regimen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Reduction of Systolic BP, diastolic BP, mean BP and pulse pressure levels will be used to compare sequential nephron blockade versus dual blockade of the renin-angiotensin-aldosterone system plus bisoprolol | Twenty weeks
  Systolic BP (mmHg), Diastolic BP (mmHg), Mean BP (mmHg) and Pulse Pressure (mmHg)

SECONDARY OUTCOMES:
Electrolytes changes: Sodium, Potassium Chlorine after 20 weeks of treatment with sequential nephron blockade compared to dual blockade of the renin-angiotensin-aldosterone system plus bisoprolol | Twenty weeks
  Sodium (reference: 135-145 mmol/L), potassium (reference: 3.5-5.0 mmol/L) and chlorine (reference: 96-106 mEq/L)
Reduction of creatinine clearance after 20 weeks of treatment with sequential nephron blockade compared to dual blockade of the renin-angiotensin-aldosterone system plus bisoprolol | Twenty weeks
  Creatinine clearance (reference - Male: 97 to 137 mL/min and Female: 88 to 128 mL/min)
Hypotension | Twenty weeks
  Recognition of hypotension (ABPM - mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Yugar-Toledo, MD, PhD, Study Chair — Sao Jose do Rio Preto Medical School
Locations (1):
- Juan Carlos Yugar-Toledo, São José do Rio Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Knauf H, Mutschler E. Sequential nephron blockade breaks resistance to diuretics in edematous states. J Cardiovasc Pharmacol. 1997 Mar;29(3):367-72. doi: 10.1097/00005344-199703000-00010. PMID 9125675
- [Background] Blumenfeld JD, Sealey JE, Mann SJ, Bragat A, Marion R, Pecker MS, Sotelo J, August P, Pickering TG, Laragh JH. Beta-adrenergic receptor blockade as a therapeutic approach for suppressing the renin-angiotensin-aldosterone system in normotensive and hypertensive subjects. Am J Hypertens. 1999 May;12(5):451-9. doi: 10.1016/s0895-7061(99)00005-9. PMID 10342782
- [Background] Azizi M, Menard J. Combined blockade of the renin-angiotensin system with angiotensin-converting enzyme inhibitors and angiotensin II type 1 receptor antagonists. Circulation. 2004 Jun 1;109(21):2492-9. doi: 10.1161/01.CIR.0000131449.94713.AD. No abstract available. PMID 15173039
- [Background] Sociedade Brasileira de Cardiologia; Sociedade Brasileira de Hipertensao; Sociedade Brasileira de Nefrologia. [VI Brazilian Guidelines on Hypertension]. Arq Bras Cardiol. 2010 Jul;95(1 Suppl):1-51. No abstract available. Portuguese. PMID 21085756
- [Background] Sociedade Brasileira de Cardiologia (SBC); Sociedade Brasileira de Hipertensao (SBH); Sociedade Brasileira de Nefrologia (SBN). [V Guidelines for ambulatory blood pressure monitoring (ABPM) and III Guidelines for home blood pressure monitoring (HBPM)]. Arq Bras Cardiol. 2011 Sep;97(3 Suppl 3):1-24. No abstract available. Portuguese. PMID 22262107
- [Result] Kearney PM, Whelton M, Reynolds K, Whelton PK, He J. Worldwide prevalence of hypertension: a systematic review. J Hypertens. 2004 Jan;22(1):11-9. doi: 10.1097/00004872-200401000-00003. PMID 15106785
- [Result] ALLHAT Officers and Coordinators for the ALLHAT Collaborative Research Group. The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial. Major outcomes in high-risk hypertensive patients randomized to angiotensin-converting enzyme inhibitor or calcium channel blocker vs diuretic: The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). JAMA. 2002 Dec 18;288(23):2981-97. doi: 10.1001/jama.288.23.2981. PMID 12479763
- [Result] Calhoun DA, Jones D, Textor S, Goff DC, Murphy TP, Toto RD, White A, Cushman WC, White W, Sica D, Ferdinand K, Giles TD, Falkner B, Carey RM. Resistant hypertension: diagnosis, evaluation, and treatment. A scientific statement from the American Heart Association Professional Education Committee of the Council for High Blood Pressure Research. Hypertension. 2008 Jun;51(6):1403-19. doi: 10.1161/HYPERTENSIONAHA.108.189141. Epub 2008 Apr 7. PMID 18391085
- [Result] Alessi A, Brandao AA, Coca A, Cordeiro AC, Nogueira AR, Diogenes de Magalhaes F, Amodeo C, Saad Rodrigues CI, Calhoun DA, Barbosa Coelho E, Pimenta E, Muxfeldt E, Consolin-Colombo FM, Salles G, Rosito G, Moreno H Jr, Martin JF, Yugar JC, Aparecido Bortolotto L, Nazario Scala LC, Goncalves de Sousa M, Gomes MA, Malachias MB, Gus M, Passarelli O Jr, Jardim PC, Toscano PR, Sanchez RA, Dischinger Miranda R, Povoa R, Barroso WK. First Brazilian position on resistant hypertension. Arq Bras Cardiol. 2012 Jul;99(1):576-85. doi: 10.1590/s0066-782x2012000700002. No abstract available. English, Portuguese. PMID 22948302
- [Result] Persell SD. Prevalence of resistant hypertension in the United States, 2003-2008. Hypertension. 2011 Jun;57(6):1076-80. doi: 10.1161/HYPERTENSIONAHA.111.170308. Epub 2011 Apr 18. PMID 21502568
- [Result] de la Sierra A, Segura J, Banegas JR, Gorostidi M, de la Cruz JJ, Armario P, Oliveras A, Ruilope LM. Clinical features of 8295 patients with resistant hypertension classified on the basis of ambulatory blood pressure monitoring. Hypertension. 2011 May;57(5):898-902. doi: 10.1161/HYPERTENSIONAHA.110.168948. Epub 2011 Mar 28. PMID 21444835
- [Result] Faselis C, Doumas M, Papademetriou V. Common secondary causes of resistant hypertension and rational for treatment. Int J Hypertens. 2011 Mar 2;2011:236239. doi: 10.4061/2011/236239. PMID 21423678
- [Result] Alvarez-Alvarez B, Abad-Cardiel M, Fernandez-Cruz A, Martell-Claros N. Management of resistant arterial hypertension: role of spironolactone versus double blockade of the renin-angiotensin-aldosterone system. J Hypertens. 2010 Nov;28(11):2329-35. doi: 10.1097/HJH.0b013e32833d4c99. PMID 20651602
- [Derived] Yugar-Toledo JC, Minari TP, de Mello PG, do Espirito Santo Cestario E, de Azevedo Rubio T, da Costa LMC, Yugar LBT, Sedenho-Prado LG, Tacito LHB, Cosenso-Martin LN, Fattori A, Pisani LP, Vilela-Martin JF, Moreno H. Effects of different antihypertensive drug classes on central and ambulatory blood pressure in resistant hypertension: A randomized clinical trial. Br J Clin Pharmacol. 2026 Jan;92(1):186-197. doi: 10.1002/bcp.70249. Epub 2025 Aug 26. PMID 40859651
- [Derived] Cestario EDES, Fernandes LAB, Giollo-Junior LT, Uyemura JRR, Matarucco CSS, Landim MIP, Cosenso-Martin LN, Tacito LHB, Moreno H Jr, Vilela-Martin JF, Yugar-Toledo JC. Resistant Hypertension On Treatment (ResHypOT): sequential nephron blockade compared to dual blockade of the renin-angiotensin-aldosterone system plus bisoprolol in the treatment of resistant arterial hypertension - study protocol for a randomized controlled trial. Trials. 2018 Feb 12;19(1):101. doi: 10.1186/s13063-017-2343-3. PMID 29433578